CLINICAL TRIAL: NCT00161707
Title: Phase I Safety Investigation of an Aerosolized, Recombinant Alpha 1-Antitrypsin in Subjects With Alpha 1-Antitrypsin Deficiency
Brief Title: Safety Study of an Aerosolized, Recombinant Alpha 1-Antitrypsin in Subjects With Alpha 1-Antitrypsin Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Arriva Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 410103
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

INTERVENTIONS:
Drug: Aerosolized, Recombinant Alpha 1-Antitrypsin

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to evaluate the short-term safety of inhaled recombinant alpha 1-antitrypsin (rAAT) in subjects with alpha 1-antitrypsin deficiency. The subjects are randomized to receive placebo or one of 4 doses of rAAT. The 4 doses are tested in a consecutive manner from lowest to highest.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Endogenous plasma AAT levels < 11 µM (< 80 mg/dL)
* Baseline forced expiratory volume at one second (FEV1) that is >= 50% of predicted, measured 30 minutes after a short-acting inhaled bronchodilator
* Baseline arterial oxygen percent saturation (SaO2) within the normal limits for the individual study site
* For subjects receiving an inhaled corticosteroid, β-2 agonist (eg, albuterol via metered dose inhaler [MDI]) or anticholinergic bronchodilator (eg, ipratropium bromide), treatment on a stable dose for at least 14 days prior to randomization
* If female of childbearing potential, negative urine pregnancy test within 3 days prior to randomization and agreement to employ adequate birth control measures
* No clinically significant abnormalities detected on a 12-lead electrocardiogram (ECG) performed no more than 7 days prior to randomization
* Baseline laboratory results, obtained no more than 7 days prior to randomization, meeting the following criteria:
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) <= 2 times upper limit of normal range (ULN)
* Serum total bilirubin <= 2 times ULN
* < 2+ proteinuria on urine dipstick
* Serum creatinine <= 1.5 times ULN
* Absolute neutrophil count >= 1500 cells/mm3
* Hemoglobin >= 10.0 g/dL
* Platelet count >= 100,000/mm3
* Signed informed consent

Exclusion Criteria:

* Clinically significant pulmonary impairment, other than emphysema and/or chronic bronchitis
* Clinically significant cardiac, hemostatic, or neurologic impairment, or other significant medical condition that, in the opinion of the investigator, would affect subject safety or compliance
* Psychiatric or cognitive disturbance or illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance
* Acute exacerbation of emphysema (as defined in Section 8.5.10) within 28 days prior to randomization
* Pregnancy or lactation
* Known history of allergy to yeast products
* Medical history precluding the use of epinephrine or other rescue medication for treatment of anaphylaxis
* Use of antihistamines within 7 days prior to randomization
* Use of oral steroids, beta-blockers, or tricyclic antidepressants within 28 days prior to randomization
* Use of another investigational drug or investigational device within 28 days prior to randomization
* Any upper or lower respiratory infection within 28 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-01-07 (Actual); Primary Completion 2003-10-01 (Actual); Study Completion 2003-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop antibodies to Recombinant Alpha 1-Antitrypsin (rAAT) | 6 weeks after the first inhalation of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - National Jewish Medical and Research Center, Denver, Colorado
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Cleveland Clinic Foundation, Department of Pulmonary and Critical Care Medicine, Cleveland, Ohio
  - The University of Texas Health Science Center at Tyler, Tyler, Texas